CLINICAL TRIAL: NCT06842901
Title: Feasibility Study on Portable Rehabilitation (PoRi) Device in Hand Spasticity
Brief Title: Feasibility Study on PoRi Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2000039568
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hand Spasticity

STUDY DESIGN:
Intervention Model Description: The study population only includes participants who present for follow up management of hand spasticity at the Yale New Haven Hospital's Physical Medicine and Rehabilitation (PM&R) outpatient clinic or who are admitted to the Yale New Haven Hospital's Inpatient Rehabilitation Unit (IRU).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hand Spasticity (Experimental): Each participant will have a single 20 minute session, during which the device will extend and flex finger muscles. Each participant's duration will be approximately 1 hour during clinic, including time to address any further questions, to calibrate the device, and data collection.
  Interventions: Device: Portable Rehabilitation (PoRi) device

INTERVENTIONS:
Device: Portable Rehabilitation (PoRi) device — Once the calibration is complete, the device moves the fingers to close and open the hand for a total of 20 minutes.

SUMMARY:
This study is a feasibility study of a new device that moves the hand of patients with spasticity to reduce hand muscle tone. The device's ability to improve spasticity before and after a 20-minute session with the device at Yale New Haven Hospital's outpatient clinic of Physical Medicine & Rehabilitation, or the Inpatient Rehabilitation Unit.

DETAILED DESCRIPTION:
Each patient will participate in a single 20 minute session, during which the device will extend and flex finger muscles. Each participant's duration will be approximately 1 hour during clinic, including time to address any further questions, to calibrate the device, and to measure the Modified Ashworth Score (MAS) before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Modified Ashworth Scale (MAS) score of at least 1
* Participants with paralysis or motor function problems of the fingers of one or both hands.

Exclusion Criteria:

* Minors (below age 18)
* Vulnerable populations
* Inability of fingers and wrist to stretch to neutral during passive range of motion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Feasibility assessed using the change in Modified Ashworth Scale (MAS) score | immediately prior to intervention session and immediately following 20 minute intervention session
  Muscle tone is rated on a 6-point scale (0, 1, 1+, 2, 3, 4) with higher scores indicating greater spasticity.

SECONDARY OUTCOMES:
Device usability and accessibility survey | immediately following 20 minute intervention session
  Device usability and accessibility will be evaluated through a patient and researcher survey.

CONTACTS AND LOCATIONS:
Overall Officials: Necolle Morgado-Vega, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - , Yale New Haven Hospital's Physical Medicine & Rehabilitation (PM&R) outpatient clinic, New Haven, Connecticut
  - Yale New Haven Hospital's Inpatient Rehabilitation Unit, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No